CLINICAL TRIAL: NCT01461876
Title: Changes in Overweight/Obesity Status, hsCRP, and D-dimer in HIV-infected Patients After 12 Months of Initial Antiretroviral Treatment
Brief Title: Obesity in HIV After Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00020911
Record Dates: First submitted 2011-10-10; First posted 2011-10-28 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2014-05

CONDITIONS: HIV; AIDS; Obesity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Obesity | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — These samples represent residual plasma retained after clinical testing (HIV RNA PCR) has been completed. Since the samples were obtained as part of routine clinical care, they are part of the HIV samples repository at Duke University Medical Center.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-infected cohort
  Interventions: Drug: antiretroviral therapy
- HIV-uninfected control group

INTERVENTIONS:
Drug: antiretroviral therapy — Standard of care antiretroviral therapy
  Groups: HIV-infected cohort

SUMMARY:
This is a retrospective longitudinal study that evaluates the prevalence and incidence of overweight/obesity within an HIV-infected population before and after 12 and 24 months of a stable antiretroviral therapy (ART). The study group will be compared to the weight of a healthy, matched population that is not infected with HIV. The primary hypothesis states that the proportion of HIV-infected persons newly classified as overweight/obese will increase by ≥20% after 12 months of initial ART, and this incidence will be greater than that of a matched HIV-uninfected control population. The effect of immune function variables, such as CD4, HIV viral load, and ART regimen on weight will be analyzed. In addition, the study will analyze the effect of weight and immune function markers on the inflammatory markers, high sensitivity C-reactive protein (hsCRP) and D-dimer. An HIV samples repository will be used for specimens to be assayed for hsCRP and D-dimer.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for HIV-infected cohort:

  1. Treatment-naive at study entry;
  2. Subjects will need to remain on ART for 12 months as initiated with substitution allowed for toxicity management within the same class of drug;
  3. Subjects within this group that remain on ART for an additional 12 months (total 24 months) as initiated with substitution allowed for toxicity management within the same class of drug will continue to be followed longitudinally for the 24 month period;
  4. Availability of repository samples.

     Inclusion Criteria for Control Cohort:

     Followed in the Duke Primary Care Clinics during the years of inclusion with available data on weight, race and gender.

     Exclusion Criteria:

Exclusion Criteria for HIV-infected cohort:

1. Pregnancy during period of observation or within 6 months of study entry;
2. Malignancy (other than squamous or basal cell carcinomas of the skin);
3. Newly diagnosed thyroid disorder within 6 months of study entry;
4. Use of megace or marinol;
5. Long-term use of glucocorticoids (greater than 1 month of prednisone 5mg or higher or an equivalent dose of another glucocorticoid);
6. Use of androgenic steroids;
7. History of diabetes or use of glucose-lowering agents;
8. Use of the following psychiatric or anticonvulsant agents- thioridazine, olanzapine (zyprexa), clozapine (clozaril), quetiapine (seroquel), risperidone (risperdal), lithium, remeron, paxil, valproate, carbamazepine, gabapentin;
9. Concurrent treatment for hepatitis C infection;
10. Diagnosis of a new opportunistic infection (OI) as defined by the CDC during the 1st 12 months of ART.22 OIs include the following: PCP, toxoplasmosis, MAC, histoplasmosis, candidiasis, cryptococcus, coccidiodes, CMV, cryptosporidium, microsporidiosis, tuberculosis, bartonellosis, herpes simplex virus, HHV-8, human papillomavirus;
11. Diagnosis of congestive heart failure and receiving diuretic therapy;
12. End stage renal disease.

Exclusion Criteria for Control Cohort:

1. Pregnancy during period of observation or within 6 months of study entry;
2. Malignancy (other than squamous or basal cell carcinomas of the skin);
3. Newly diagnosed thyroid disorder within 6 months of study entry;
4. Long-term use of glucocorticoids (greater than 1 month of prednisone 5mg or higher or an equivalent dose of another glucocorticoid);
5. Use of androgenic steroids;
6. History of diabetes or use of glucose-lowering agents;
7. Use of the following psychiatric or anticonvulsant agents- thioridazine, olanzapine (zyprexa), clozapine (clozaril), quetiapine (seroquel), risperidone (risperdal), lithium, remeron, paxil, valproate, carbamazepine, gabapentin;
8. Treatment for hepatitis C infection during observation period;
9. Diagnosis of congestive heart failure and receiving diuretic therapy;
10. End stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (≥ 18 years of age) infected with HIV-1 treated in the Infectious Disease Clinic at Duke University Medical Center between 3/1/98 to 3/1/08 who meet eligibility criteria.
  Adult subjects (≥ 18 years of age), followed in primary care clinics within the Duke Health System between 3/1/98 to 3/1/08, who meet eligibility criteria. Control subjects must have data for weight 12 months after baseline visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in BMI from baseline after 12 months of initial antiretroviral therapy | 12 months

SECONDARY OUTCOMES:
Change in the inflammatory marker, high-sensitivity C-reactive protein, from baseline after 12 months of antiretroviral therapy | 12 Months
Change in the prothrombotic marker, D-dimer, from baseline after 12 months of initial antiretroviral therapy | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Lakey, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States